CLINICAL TRIAL: NCT02340299
Title: Nasal High Frequency Oscillation Ventilation Versus Nasal Continuous Positive Airway Pressure to Reduce Post-extubation pCO2 in Very Low Birth Weight Infants: a Randomized Controlled Trial
Brief Title: Nasal HFOV Versus Nasal CPAP to Reduce Post-extubation pCO2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Christoph Czernik, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2/011/12
Record Dates: First submitted 2015-01-10; First posted 2015-01-16 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Distress Syndrome, Newborn; Respiratory Tract Diseases
Keywords: High Frequency Oscillation Ventilation; Nasal Continuous Positive Airway Pressure; Airway Extubation; Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Tract Diseases; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nHFOV (Experimental): Immediately after extubation, nHFOV is provided via binasal prongs. Ventilator settings: Frequency set at 10 Hz, I:E ratio 33:66, amplitude 20 cm H2O, Pmean 8 cm H2O, flow 7 l/min. Set FiO2 to maintain SpO2 at 90-94%.
  The weaning process is left to the discretion of the attending physician. Maximum amplitude 30 cm H2O, minimum frequency 9 Hz, maximum Pmean 8 cm H2O.
  For infants in the nHFOV-group who "fail" nHFOV (see definition below), but do not need immediate reintubation, a non-invasive "Rescue-Treatment" may be provided. The decision to attempt "Rescue-Treatment", the mode of respiratory support and the ventilator settings used are at the discretion of the attending clinician.
  Interventions: Device: nHFOV
- nCPAP (Active Comparator): Immediately after extubation, nCPAP is provided via binasal prongs. Ventilator settings: CPAP level set at 8 cm H2O, flow 7 l/min. Set FiO2 to maintain SpO2 at 90-94%.
  The weaning process is left to the discretion of the attending physician. Maximum CPAP level 8 cm H2O, maximum flow 8 l/min.
  For infants in the nCPAP-group who "fail" nCPAP (see definition below), but do not need immediate reintubation, "Rescue-nHFOV" via binasal prongs may be provided. The decision to attempt "Rescue-nHFOV" and the ventilator settings used are at the discretion of the attending clinician.
  Interventions: Device: nCPAP

INTERVENTIONS:
Device: nHFOV — Extubation to ventilator-derived nHFOV using binasal prongs
  Arms: nHFOV
Device: nCPAP — Extubation to ventilator-derived nCPAP using binasal prongs
  Arms: nCPAP

SUMMARY:
To investigate whether nasal high frequency oscillation ventilation (nHFOV) immediately after extubation reduces the arterial partial pressure of carbon dioxide (paCO2) at 72 hours after extubation in comparison with nasal continuous positive airway pressure (nCPAP) in very low birth weight infants (VLBWs).

DETAILED DESCRIPTION:
Randomized controlled clinical trial comparing nHFOV vs nCPAP immediately after extubation of VLBW infants.

Intervention and treatment protocol as described for the two study arms.

Definition of treatment failure (infant meets at least one criterion):

* Sustained pCO2 >80 mmHg and pH <7.20 confirmed by arterial or capillary blood gas analysis in spite of optimized non-invasive respiratory support with maximum settings as defined above.
* Fraction of inspired oxygen (FiO2) >0.6 to maintain peripheral oxygen saturation as measured by pulse oximetry (SpO2) at 90-94% in spite of optimized non-invasive respiratory support with maximum settings as defined above.
* Reintubation (study patients may be intubated at any time, due to clinical considerations, with or without reaching another criterion of "treatment failure").

Sample size:

Assuming a variability of the paCO2 as previously reported for difficult-to-wean preterm infants in our unit (Czernik C, J Matern Fetal Neonatal Med 2012) and a treatment failure rate of 22% within 72 hours after extubation, we calculated a sample size of 34 patients in each study arm to detect a difference in the paCO2 of 7 mmHg, using a two-sided significance of 0.05 and a power of 0.8.

Randomization:

Sequence generation by an independent statistician and a study nurse. Block randomization using at least two different block sizes. Allocation concealment using sequentially numbered opaque sealed envelopes.

Data monitoring:

By an independent statistician.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <32+0 weeks
* Birth weight <1500 g
* Received mechanical ventilation via an endotracheal tube for ≥120 h
* Caffeine treatment according to unit guidelines
* paCO2 <65 mmHg with pH >7.2
* FiO2 25-40% to maintain SpO2 at 90-94%.
* Time-cycled, pressure-controlled ventilation: PIP ≤22 cm H2O, PEEP ≤6 cm H2O; Volume guarantee ventilation: Working Ppeak ≤22 cm H2O, PEEP ≤6 cm H2O; High frequency oscillation ventilation: Pmean ≤12 cm H2O, Amplitude ≤30 cm H2O
* Decision of the attending clinician to extubate

Exclusion Criteria:

* Major congenital malformation requiring surgery
* Duct-dependent congenital heart disease
* Neuromuscular disease
* Participation in another randomized controlled trial
* Death before reaching the eligibility criteria
* Hydrocortisone treatment at the time of enrolment
* Chronological age >28 days

Ages: 5 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Czernik, MD PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Dpt. of Neonatology, Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Fischer HS, Buhrer C, Czernik C. Hazards to avoid in future neonatal studies of nasal high-frequency oscillatory ventilation: lessons from an early terminated trial. BMC Res Notes. 2019 Apr 25;12(1):237. doi: 10.1186/s13104-019-4268-2. PMID 31023363

RESULTS

PARTICIPANT FLOW:
Groups:
- nHFOV: Immediately after extubation, nHFOV is provided via binasal prongs. Ventilator settings: Frequency set at 10 Hz, I:E ratio 33:66, amplitude 20 cm H2O, Pmean 8 cm H2O, flow 7 l/min. Set FiO2 to maintain SpO2 at 90-94%.
  The weaning process is left to the discretion of the attending physician. Maximum amplitude 30 cm H2O, minimum frequency 9 Hz, maximum Pmean 8 cm H2O.
  For infants in the nHFOV-group who "fail" nHFOV (see definition below), but do not need immediate reintubation, a non-invasive "Rescue-Treatment" may be provided. The decision to attempt "Rescue-Treatment", the mode of respiratory support and the ventilator settings used are at the discretion of the attending clinician.
  nHFOV: Extubation to ventilator-derived nHFOV using binasal prongs
- nCPAP: Immediately after extubation, nCPAP is provided via binasal prongs. Ventilator settings: CPAP level set at 8 cm H2O, flow 7 l/min. Set FiO2 to maintain SpO2 at 90-94%.
  The weaning process is left to the discretion of the attending physician. Maximum CPAP level 8 cm H2O, maximum flow 8 l/min.
  For infants in the nCPAP-group who "fail" nCPAP (see definition below), but do not need immediate reintubation, "Rescue-nHFOV" via binasal prongs may be provided. The decision to attempt "Rescue-nHFOV" and the ventilator settings used are at the discretion of the attending clinician.
  nCPAP: Extubation to ventilator-derived nCPAP using binasal prongs
Period: Overall Study
Arm/Group | nHFOV | nCPAP
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | nHFOV | nCPAP | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: days] | 19 [15 to 28] | 16 [13 to 19] | 17.5 [13 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: paCO2 at 72 h After Extubation
Description: Partial pressure of arterial carbon dioxide assessed between 64 and 80 hours, and on average 72 hours.
Time Frame: 64 h to 80 h
Population: In patients that were reintubated within 72 h, the primary outcome, paCO2 72 h after extubation, could not be assessed. In the nCPAP group, all patients had to be reintubated within 72 h. The primary outcome, paCO2 72 h after extubation, could therefore only be assessed in the nHFOV group.
Measure: Median (Full Range); unit: mmHg
Arm/Group | nHFOV | nCPAP
Number analyzed (Participants) | 2 | 0
mmHg | 65.5 [52 to 79] |

2. Secondary Outcome: pH at 2 h After Extubation
Time Frame: within the first 6 h after extubation
Reporting Status: Not Posted

3. Secondary Outcome: paO2 at 2 h After Extubation
Time Frame: within the first 6 h after extubation
Reporting Status: Not Posted

4. Secondary Outcome: paCO2 at 2 h After Extubation
Time Frame: within the first 6 h after extubation
Reporting Status: Not Posted

5. Secondary Outcome: Base Excess at 2 h After Extubation
Time Frame: within the first 6 h after extubation
Reporting Status: Not Posted

6. Secondary Outcome: pH at 72 h After Extubation
Time Frame: 64-80 h after extubation
Reporting Status: Not Posted

7. Secondary Outcome: paO2 at 72 h After Extubation
Time Frame: 64-80 h after extubation
Reporting Status: Not Posted

8. Secondary Outcome: Base Excess at 72 h After Extubation
Time Frame: 64-80 h after extubation
Reporting Status: Not Posted

9. Secondary Outcome: Successful Extubation
Description: Defined as the number of patients breathing spontaneously in their assigned treatment group for ≥72h without reaching the criterion of "treatment failure"
Time Frame: 72 h after extubation
Reporting Status: Not Posted

10. Secondary Outcome: Treatment Failure
Description: Defined as the number of patients reaching the criterion of "treatment failure"
Time Frame: within 7 days after extubation
Reporting Status: Not Posted

11. Secondary Outcome: Reintubation
Description: Defined as the number of patients being reintubated
Time Frame: within 7 days after extubation
Reporting Status: Not Posted

12. Secondary Outcome: Highly Viscous Secretions
Description: Defined as the documented number of episodes of airway obstruction due to highly viscous secretions per patient
Time Frame: within 72 hours after extubation
Reporting Status: Not Posted

13. Secondary Outcome: Other Adverse Effects
Description: Incidences of the following adverse effects: Intraventricular hemorrhage III°-IV° (Papile), surgical necrotizing enterocolitis, pneumothorax, pulmonary interstitial emphysema, persistent ductus arteriosus requiring surgical closure, retinopathy of prematurity requiring laser treatment and/or injection of bevacizumab, death or moderate to severe bronchopulmonary dysplasia (Jobe) at 36 weeks' gestational age, periventricular leukomalacia
Time Frame: until discharge
Reporting Status: Not Posted

14. Secondary Outcome: Duration of Respiratory Support
Description: Total duration of mechanical ventilation, total duration of supplemental oxygen, number of infants discharged with home oxygen
Time Frame: until discharge
Reporting Status: Not Posted

15. Other Pre Specified Outcome: pH at 2 h After Switch to "Rescue Treatment"
Time Frame: within the first 6 h after switch to "rescue treatment"
Reporting Status: Not Posted

16. Other Pre Specified Outcome: paO2 at 2 h After Switch to "Rescue Treatment"
Time Frame: within the first 6 h after switch to "rescue treatment"
Reporting Status: Not Posted

17. Other Pre Specified Outcome: paCO2 at 2 h After Switch to "Rescue Treatment"
Time Frame: within the first 6 h after switch to "rescue treatment"
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Base Excess at 2 h After Switch to "Rescue Treatment"
Time Frame: within the first 6 h after switch to "rescue treatment"
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Successful Rescue
Description: Defined as spontaneous breathing for ≥72h after starting "rescue" therapy, without reaching the criterion of "treatment failure"
Time Frame: 72 h after switch to "rescue" treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected until discharge from the neonatal unit. Patients were discharged approximately at 3 months of age.
Arm/Group | nHFOV | nCPAP
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/4 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nHFOV (N=4) | nCPAP (N=2)
Highly viscous secretions (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT02340299/Prot_SAP_000.pdf